CLINICAL TRIAL: NCT02410356
Title: A Phase 3, Multicenter, Randomized, Open-Label, Comparator-Controlled Study to Assess Safety and Tolerability of Weekly TV-1106 Compared to Daily rhGH (Genotropin(R)) in Adults With Growth Hormone-Deficiency
Brief Title: Study to Assess Safety and Tolerability in Adults With Growth Hormone-Deficiency (GHD)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business decision
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TV1106-IMM-30022
Record Dates: First submitted 2015-03-30; First posted 2015-04-07 (Estimated); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — albusomatropin; Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TV-1106 (Experimental): TV-1106 to be injected once weekly.
  Interventions: Drug: TV-1106
- dGH (Active Comparator): dGH to be given as daily injections.
  Interventions: Drug: dGH

INTERVENTIONS:
Drug: TV-1106 — The volume necessary to provide the required weekly dose will be calculated by the investigator; dose will be adjusted for IGF-I in the normal range.
  Other Names: rhGH
  Arms: TV-1106
Drug: dGH — The dose levels of dGH will be the same as the stable rhGH dose taken prior to the study.
  Other Names: rhGH; Somatropin
  Arms: dGH

SUMMARY:
This study assesses the safety and tolerability of weekly TV-1106 compared to daily rhGH in adults with GHD who have previously been treated with rhGH.

ELIGIBILITY:
Inclusion Criteria:

* males and females 18 years of age or over
* diagnosis of adult GHD for at least 6 months, or patients who have hypopituitarism from surgical resection
* treated with a stable dose of daily rhGH for at least 3 months prior to screening
* stable, adequate doses of replacement hormones (adrenal, thyroid, estrogen, testosterone, vasopressin) for at least 3 months prior to screening

  * Other criteria apply, please contact the investigator for more information

Exclusion Criteria:

* patients with acute or chronic conditions or diseases that could confound results of the study or put the patient at undue risk as determined by the investigator
* Presence of contraindications to rhGH treatment
* patients who have participated in another clinical trial with a new chemical/biological entity within 3 months of screening
* patients with known active malignancy (excluding surgically removed basal cell carcinoma or carcinoma in situ of cervix) d. patients with a previously treated pituitary tumor with evidence of tumor progression in the past year
* patients with a new diagnosis of pituitary adenoma or other intracranial tumor within 12 months of screening
* presence of Prader-Willi syndrome, Turner's syndrome, untreated adrenal insufficiency, active acromegaly in the past 5 years, or active Cushing's syndrome in the past year.
* patients with type 1 diabetes mellitus oror poorly controlled type 2 diabetes mellitus as indicated by a glycated hemoglobin (HbA1c) ≥8%
* patients using weight reducing agents or appetite suppressants

  * Other criteria apply, please contact the investigator for more information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-04-30 (Actual); Primary Completion 2016-02-29 (Actual); Study Completion 2016-04-30 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with adverse events | 48 weeks
  Safety of TV-1106 compared to reference drug

SECONDARY OUTCOMES:
Change from baseline in Insulin-like Growth Factor 1 Standard Deviation Score | Baseline, Weeks: 4, 8, 12, 16, 24, 36, 48

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (50):
- United States (32):
  - Teva Investigational Site 13137, Artesia, California
  - Teva Investigational Site 13166, Fountain Valley, California
  - Teva Investigational Site 13165, Lakewood, California
  - Teva Investigational Site 13155, Denver, Colorado
  - Teva Investigational Site 13158, Newark, Delaware
  - Teva Investigational Site 13162, Fort Lauderdale, Florida
  - Teva Investigational Site 13136, Homestead, Florida
  - Teva Investigational Site 13138, Miami, Florida
  - Teva Investigational Site 13152, Miami, Florida
  - Teva Investigational Site 13161, Miami, Florida
  - Teva Investigational Site 13500, Miami, Florida
  - Teva Investigational Site 13503, Miami, Florida
  - Teva Investigational Site 13148, Miami Lakes, Florida
  - Teva Investigational Site 13134, Pembroke Pines, Florida
  - Teva Investigational Site 13129, West Palm Beach, Florida
  - Teva Investigational Site 13135, Detroit, Michigan
  - Teva Investigational Site 13146, Henderson, Nevada
  - Teva Investigational Site 13147, Las Vegas, Nevada
  - Teva Investigational Site 13143, Brooklyn, New York
  - Teva Investigational Site 13502, New York, New York
  - Teva Investigational Site 13140, New York, New York
  - Teva Investigational Site 13128, Asheville, North Carolina
  - Teva Investigational Site 13142, Pittsburgh, Pennsylvania
  - Teva Investigational Site 13144, Arlington, Texas
  - Teva Investigational Site 13163, Dallas, Texas
  - Teva Investigational Site 13130, Houston, Texas
  - Teva Investigational Site 13141, Houston, Texas
  - Teva Investigational Site 13154, Houston, Texas
  - Teva Investigational Site 13159, Norfolk, Virginia
  - Teva Investigational Site 13504, Federal Way, Washington
  - Teva Investigational Site 13164, Seattle, Washington
  - Teva Investigational Site 13157, Tacoma, Washington
- Teva Investigational Site 33035, Linz, Austria
- Czechia (3):
  - Teva Investigational Site 54118, Brno
  - Teva Investigational Site 54119, Moravskoslezsky
  - Teva Investigational Site 54116, Plzensky
- Greece (3):
  - Teva Investigational Site 63059, Athens
  - Teva Investigational Site 63058, Chaïdári
  - Teva Investigational Site 63060, Ioannina
- Hungary (6):
  - Teva Investigational Site 51202, Budapest
  - Teva Investigational Site 51206, Budapest
  - Teva Investigational Site 51205, Debrecen
  - Teva Investigational Site 51204, Pécs
  - Teva Investigational Site 51208, Szeged
  - Teva Investigational Site 51207, Szolnok
- Teva Investigational Site 30129, Brescia, Italy
- Teva Investigational Site 62041, Ľubochňa, Slovakia
- Spain (3):
  - Teva Investigational Site 31129, Badalona
  - Teva Investigational Site 31121, Córdoba
  - Teva Investigational Site 31125, Madrid